CLINICAL TRIAL: NCT00669045
Title: A Phase IV, Prospective, Observational Study of TNKase in Patients Enrolled in the National Registry of Myocardial Infarction 4 and 5 (POST)
Brief Title: An Observational Study of TNKase in Patients Enrolled in the National Registry of Myocardial Infarction 4 and 5 (POST)
Status: Completed | Type: Observational
Sponsor: Genentech, Inc. (Industry)
Other Study IDs: N2224n
Record Dates: First submitted 2008-04-27; First posted 2008-04-29 (Estimated); Last update posted 2017-02-15 (Actual); Status verified 2017-02

CONDITIONS: Acute Myocardial Infarction
Keywords: TNKase; AMI

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective

SUMMARY:
The POST study comprised patients whose data were entered into the NRMI 4 and 5 databases. NRMI is a prospective, observational study of patients presenting with AMI in the United States. NRMI was launched in 1990 and to date has enrolled more than 2.5 million AMI patients. More than 1,700 hospitals have participated in NRMI during the last 16 years. The NRMI 4 and 5 substudies were sponsored by Genentech and collected data on approximately 160,000 AMI patients (both ST elevation and non-ST-elevation MI) hospitalized in the United States each year. This corresponds to approximately 18% of the AMI patients in the United States.

ELIGIBILITY:
Inclusion Criteria:

* Presence of LBBB or ST-segment elevation (new or of unknown duration)
* ICD-9-CM discharge code of 410.X1
* Treatment with one of the following regimens: TNKase; Other thrombolytic regimens; No initial reperfusion

Exclusion Criteria:

* Patients who were transferred out of the facility
* Patients with pending data clarification forms on fields related to study variables

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 253668 (Actual)
Dates: Start 2000-09-01 (Actual); Primary Completion 2006-03-31 (Actual); Study Completion 2006-03-31 (Actual)